CLINICAL TRIAL: NCT02230215
Title: Assessment of Conventional and Patient-specific Instrumentation in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Orthopaedic Foundation (Other); Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Douglas Naudie, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 105453
Record Dates: First submitted 2014-08-19; First posted 2014-09-03 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis
Keywords: Total Knee Replacement; Visionaire
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient-Specific Instrumentation (Experimental): Patients to have a total knee replacement surgery completed using Patient-Specific Instrumentation
  Interventions: Device: Total Knee Arthroplasty with use of Visionaire Patient-Specific Instrumentation
- Traditional Instrumentation (No Intervention): Patients to have a total knee replacement surgery done using traditional instrumentation.

INTERVENTIONS:
Device: Total Knee Arthroplasty with use of Visionaire Patient-Specific Instrumentation — The manufacturing of a patient-specific instrument to be used by the orthopaedic surgeon during the knee replacement surgery.
  Other Names: Visionaire Patient Specific Instrumentation
  Arms: Patient-Specific Instrumentation

SUMMARY:
This study will use a special type of x-ray called radiostereometric analysis (RSA) imaging to determine whether patient-specific instrumentation for total knee arthroplasty (replacement) has an effect on implant loosening compared to conventional instrumentation. Secondary objectives will include assessment of post-operative implant alignment, patient satisfaction, operative time and surgical instrument use, cost, and environmental impact.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial which will enroll 50 patients undergoing total knee replacement surgery. All study patients will undergo an MRI prior to surgery. Half (25)of these patients will be randomized to have their MRI used to develop a patient-specific instrument to be used during their surgery. The other half (25) will have conventional instrumentation (CI) used for their knee replacement surgery.

All patients will have the same type of knee implant used for their total knee replacement (Genesis II posterior stabilized (Smith & Nephew).

Patients will not know which group they have been randomized to. For patients randomized into the patient-specific randomization group, If the surgeon is not happy with the patient-specific instrumentation, they have the option to switch to conventional instrumentation at any time during the surgery.

• Length of operation, number of instruments used, amount of OR room waste and number and type of adjustments to the patient specific instrumentation will be tracked.

During the surgery, all patients in the study will have tantalum marker beads placed in the bone surrounding their knee replacement. These beads will be used as markers to measure implant fixation over the next two years. All patients will undergo a special type of x-ray imaging called RSA imaging to quantify implant fixation over time.

RSA examinations will occur at 6 weeks, 3 months, 6 months, 1 year, and 2 years at the Robart's Research Institute after their standard of care visit with orthopaedic surgeon.

Model based RSA software used to measure motion of implant components relative to bone markers.

All patients will complete our standard outcome measures in the form of surveys completed at their follow-up visits after surgery. •

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary total knee replacement surgery
* No previous knee hardware (ie.Uni-Knees, or high tibial osteotomy)
* BMI < 40
* Study patients should live within 100 km of our facility to ensure availability for follow-up

Exclusion Criteria:

* Pregnancy or considering pregnancy
* BMI > 40
* Unable to undergo MRI screening

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Evaluating the Change in Implant Fixation assessed using RSA imaging | 2 weeks, 6 weeks, 3 months 6 months, 1 year, 2 years
  Model based RSA will be used to measure the migration of the implant components relative to the bone between all time points.

SECONDARY OUTCOMES:
Patient Outcomes including Satisfaction | Preoperatively, 1 year, 2 year
  Patient reported outcome measures provide important insight into how well total knee replacement performs from the patient's perspective. We will obtain patient surveys using four common, validated outcome measures: Knee Society Score, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Short Form 12 Health Survey (SF-12), and University of California, Los Angeles (UCLA) Activity Score

OTHER OUTCOMES:
Component Alignment | 1 year, 2 year
  Using standard 3 foot hip-to-ankle radiographs to determine radiographic alignment of the implant components and mechanical axis of the limb.
Cost | Intraoperatively
  Tracking time and instruments used per procedure and waste collected.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Naudie, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No